CLINICAL TRIAL: NCT04152850
Title: Effect of a Culturally Adapted Self-help Smartphone-based Lifestyle Intervention in Reducing Depressive and Anxiety Symptoms: A Randomized Controlled Trial
Brief Title: Self-help Lifestyle Medicine for Depression and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY009
Record Dates: First submitted 2019-11-04; First posted 2019-11-05 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Depression, Anxiety
Keywords: Depression; Anxiety; Lifestyle Medicine; Self-help
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Medicine Group (Experimental)
  Interventions: Behavioral: Lifestyle Medicine
- Waitlist Control Group (No Intervention): Participants in the waitlist control group will receive the intervention after the immediate post-treatment assessment

INTERVENTIONS:
Behavioral: Lifestyle Medicine — Lifestyle intervention with components including physical activity, diet, relaxation/mindfulness, sleep and Traditional Chinese Medicine
  Arms: Lifestyle Medicine Group

SUMMARY:
This study will examine the effects of smartphone-based lifestyle medicine (LM) for alleviating depressive and anxiety symptoms in Chinese population. Since a range of lifestyle factors are involved in the pathogenesis and progression of depression and anxiety, modifying different lifestyle factors simultaneously, for example, diet, exercise, stress and sleep which are empirically supported by previous reviews, may be effective to reduce depressive and anxiety symptoms. Traditional Chinese medicine concepts will be integrated into the app to increase the acceptability towards mental health treatment. Through this study, we aim to promote evidence-based patient care and to improve help-seeking and access to evidence-based interventions for depression and anxiety.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial on the effects of a culturally adapted self-help smartphone-based lifestyle medicine for reducing depressive and anxiety symptoms in Chinese population. Prior to all study procedures, eligible participants will be required to complete an online informed consent (with telephone support). With an estimation of 30% withdrawal, around 124 eligible participants will be randomly assigned to either smartphone-based lifestyle medicine (LM group) or the waitlist control group (WL group) in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Aged ≥ 18 years
* Have a Patient Health Questionnaire (PHQ-9) score ≥ 10 or Generalized Anxiety Disorder 7-Item Scale (GAD-7) ≥ 8
* Able to read Chinese and type in Chinese or English
* Have an Internet-enabled mobile device (iOS or Android operating system)
* Are willing to provide informed consent and comply with the trial protocol

Exclusion Criteria:

* Current involvement in psychotherapy or unstable medication for depression and/or anxiety
* Beck Depression Inventory (BDI-II) Item 9 score of at least 2 indicating a current moderate suicidal risk that requires active crisis management (referral information to professional services will be provided to those with serious suicidal risk)
* Are having unsafe conditions and are not recommended for physical activity or a change in diet by physicians
* Having major psychiatric, medical or neurocognitive disorders that make participation infeasible or interfere with the adherence to the lifestyle modification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, immediately post-treatment and 1-month post treatment
  The PHQ-9, a 9-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
Change in the Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Baseline, immediately post-treatment and 1-month post treatment
  The GAD-7, a 7-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of anxiety over the past two weeks on a 4-point scale, "0" (not at all) to "4" (nearly every day).

SECONDARY OUTCOMES:
Change in the Insomnia Severity Index (ISI) | Baseline, immediately post-treatment and 1-month post treatment
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5 point Likert scale are obtained on the perceived severity of sleep-onset, sleep maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in the Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, immediately post-treatment and 1-month post treatment
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in the Health-Promoting Lifestyle Profile (HPLP II) | Baseline, immediately post-treatment and 1-month post treatment
  The 52-item HPLPII is composed of a total scale and six subscales to measure behaviors in the theorized dimensions of health-promoting lifestyle: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management.
Change in the Sheehan Disability Scale (SDS) | Baseline, immediately post-treatment and 1-month post treatment
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
Change in the Credibility-Expectancy Questionnaire (CEQ) | Baseline, immediately post-treatment and 1-month post treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.
Change in the Food Frequency Questionnaires (FFQs) | Baseline, immediately post-treatment and 1-month post treatment
  FFQs is a 18-item scale, including drinks, plant, animal products and cigarette intake, which measures the frequency of food intake over the past three months on a 7-point scale.
Change in the International Physical Activities Questionnaire - Chinese version (IPAQ-C) (Lai et al., 2018; Macfarlane, Lee, Ho, Chan, & Chan, 2007) | Baseline, immediately post-treatment and 1-month post treatment
  Participants' sitting time, walking time and moderate and vigorous physical activity are assessed by 5 questions from the short form of the International Physical Activity Questionnaire - Chinese version. The sample questions include: "On a typical weekday in the last 7 days, how many hours per day did you typically spend sitting?"; "On a typical weekend in the last 7 days, how many hours per day did you typically spend sitting?". Participants' engagement in brief strength and stamina-enhancing activity were assessed by asking the number of days they engaged in physical activity while seated and standing in the last seven days.
Self-developed survey | Baseline
  The self-developed survey will collect information including demographic information (e.g., age, gender, level of education, working industry, relationship status, and location of residence), substance use, body mass index (BMI), rest-activity pattern, and social rhythms, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

REFERENCES:
- [Derived] Wong VW, Ho FY, Shi NK, Tong JT, Chung KF, Yeung WF, Ng CH, Oliver G, Sarris J. Smartphone-delivered multicomponent lifestyle medicine intervention for depressive symptoms: A randomized controlled trial. J Consult Clin Psychol. 2021 Dec;89(12):970-984. doi: 10.1037/ccp0000695. PMID 35025538